CLINICAL TRIAL: NCT02336074
Title: Research In Viral Eradication of HIV Reservoirs
Acronym: RIVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); University of Oxford (Other); University of Cambridge (Other); Chelsea and Westminster NHS Foundation Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Central and North West London NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCT-NAPN-24772; 2014-001425-32 (EudraCT Number)
Record Dates: First submitted 2014-10-23; First posted 2015-01-12 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: HIV
Keywords: HIV; Vaccine; Cure; Early Intervention; Infection; Primary infection; Reservoir; Vorinostat; HDAC
MeSH Terms: conditions — Infections | interventions — Antiretroviral Therapy, Highly Active; Raltegravir Potassium; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed at week 0 for the duration of the study up to post-randomisation week 18 (42 weeks in total)
  Interventions: Drug: Combination Antiretroviral Therapy (cART); Drug: Raltegravir
- Intervention (Experimental): Combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed at week 0 for the duration of the study up to post-randomisation week 18 (42 weeks in total) Plus ChAdV63.HIVconsv prime (post-randomisation week 00) and MVA.HIVconsv boost (post randomisation week 08 day 1) vaccines; followed by a 28-day course of vorinostat (10 doses in total).
  Interventions: Drug: Combination Antiretroviral Therapy (cART); Drug: Raltegravir; Drug: Vorinostat; Biological: ChAdV63.HIVconsv (ChAd); Biological: MVA.HIVconsv (MVA)

INTERVENTIONS:
Drug: Combination Antiretroviral Therapy (cART) — Likely consisting of an Nucleoside reverse-transcriptase inhibitor (NRTI) backbone i.e. Truvada plus a ritonavir-boosted protease inhibitor (PI) e.g. Darunavir + ritonavir. Prescribed at week 0 for the duration of the study.
Drug: Raltegravir — All participants will be dispensed sufficient supplies of Raltegravir to ensure they have sufficient medication to last to the next study visit. Raltegravir is supplied in marketed pack with 30 tablets per bottle.
  Other Names: Isentress
Drug: Vorinostat — Vorinostat (suberoylanilide hydroxamic acid abbreviated to SAHA) inhibits the histone deacetylases HDAC1, HDAC2, HDAC3 (Class I) and HDAC6 (Class II).
  Vorinostat is supplied as capsules containing 100mg vorinostat and the following inactive ingredients: microcrystalline cellulose, sodium croscarmellose and magnesium stearate.
  Arms: Intervention
Biological: ChAdV63.HIVconsv (ChAd) — Dosage: 5x1010vp .This dose is obtained by injecting 0.37ml of the vaccine at 1.35x1011vp/ml without dilution. This prime vaccination is administered intramuscularly (IM) into the deltoid muscle of the non-dominant arm at post-randomisation week 00.
  Arms: Intervention
Biological: MVA.HIVconsv (MVA) — Dosage: 2x108pfu Administration: This dose is obtained by injecting 0.23 ml of the vaccine IM at 8.6x108pfu/ml without dilution. This boost vaccination is administered intramuscularly (IM) into the deltoid muscle of the non-dominant arm at post-randomisation week 08 Day 1 (2 prior to start of vorinostat)
  Arms: Intervention

SUMMARY:
This study will be a two-arm prospective 1:1 randomised controlled trial comparing:

Arm A: cART preferably including raltegravir (combination ART cART - control) Arm B: cART preferably including raltegravir (cART) plus ChAdV63.HIVconsv (ChAd) prime and MVA.HIVconsv (MVA) boost vaccines; followed by a 28-day course of vorinostat (10 doses in total).

We hypothesise that this intervention in primary HIV infection will confer a significant reduction in the latent HIV reservoir when compared with cART alone.

.

DETAILED DESCRIPTION:
The study design is a two-arm, open label randomised study. Eligible participants are recruited from two participant cohorts (Cohort I - Recently diagnosed or Cohort II - Previously diagnosed with HIV). All participants receive combination ART (cART) for the duration of the intervention phase of the study (Cohort I: 42 weeks, Cohort II: 18 weeks). In patients meeting the criteria for randomisation (eligibility assessed at week 22/screening), participants will either continue cART or receive an intervention consisting of two anti-HIV vaccines separated by 8 weeks followed by 10 doses of the HDACi, vorinostat, in addition to cART. We hypothesise that the prime-boost vaccination will result in the generation of vaccine induced HIV specific CTLs that will recognise HDACi-activated cells of the HIV reservoir and destroy them. The net effect will be a greater reduction in the HIV reservoir defined as HIV total DNA in CD4+ T-cells in the cART+vaccine+HDACi compared to the cART alone. Our strategy is entirely different from previous therapeutic vaccination approaches which have been largely unsuccessful. Immunological priming to conserved HIV proteins will drive CD8+ T-lymphocyte recognition of latently-infected cells rendered immunogenic by HDACi. We anticipate that the viral antigens expressed by latently-infected cells will be unable to adapt to, or escape from, the immune response as they will be expressed directly from chromosomal DNA, avoiding the steps of the viral life-cycle that facilitate immune-driven adaptation. We have chosen a prime-boost immunisation strategy with recombinant replication-defective chimpanzee adenovirus and modified vaccinia Ankara vectors, bearing conserved HIV antigens; these products have been shown to induce high titres of HIV-specific CD8+ T-cells. In addition, these vaccines will drive immune responses against conserved regions of the virus that may be well preserved in individuals with PHI.

Primary HIV Infection (PHI) is a unique period when HIV proviral reservoir is smaller than in chronic disease, is likely to be more homogeneous than in later stage disease and hence is more susceptible to immunological elimination. This provides an opportunity to use a vaccine to re-direct HIV-specific immune responses towards genetically fragile regions in the viral proteome. Immunisation in PHI should result in potent immune responses because ART initiated in PHI preserves CD4 function and early ART-mediated viral suppression limits viral diversification, reducing the chance of immune escape. The other key reason for conducting this trial in patients treated in PHI is that, in some patients, an early sustained course of ART started very early in infection may induce a state of viral remission in which therapy can be stopped without any rebound viraemia. This has been most notably reported in the VISCONTI cohort in which 'post-treatment control' was identified in 15.6% of selected individuals.

Data from our group and others has shown that whilst there is a rapid decline in measures of total HIV DNA following ART initiation up to 6 months after seroconversion this then plateaus out to approximately 2 years after diagnosis of acute infection. Hence randomisation of individuals starting immediate ART in acute infection have comparable levels of HIV reservoirs to those who have started treatment within a similar timeframe, but have remained on suppressive therapy for up to 2 years after initiation. Furthermore, since the primary endpoint of the RIVER study design compares total HIV DNA between the two arms from randomisation to post-randomisation weeks 16 & 18 Cohorts I and II will be comparable.

We hypothesise that the combination of HDACi with immunisation in cART-suppressed PHI will significantly impact the HIV reservoir.

1. Patients in Cohort I - Recently diagnosed will receive combination antiretroviral therapy designed to reduce the plasma viral load as quickly as possible, hence the rationale for the preferred inclusion of raltegravir, an integrase inhibitor. Both cohorts will have been treated in PHI, which may restrict the size of the reservoir compared with people initiating ART in later stages of HIV infection. Cohort II - Previously diagnosed participants are screened the same as Cohort I and are maintained on ART throughout the study. The ART regimen is preferably a combination that includes raltegravir, as hypothetically, if vorinostat induced viral transcription an integrase inhibitor may protect uninfected cells. However, there is no evidence to support this hypothesis and the key inclusion criteria must be the continuation of a virally suppressive ART regimen throughout the study.
2. The prime-boost vaccination is designed to enhance the killing capacity of the cytotoxic T cells. This must be given before the HDACi in order to prime and boost a maximal HIV-specific T-cell response to recognise activated viral antigen expression on reservoir cells.
3. The HDACi is designed to cause viral transcription from latently infected cells; activate the reservoir, and in the presence of the enhanced killing capacity of the CD8+ T cells, results in killing of the cells previously harbouring latent virus, leading to further reductions in the reservoir.

This exact combined approach in treated PHI has never previously been used, we hypothesise there will be a 50% reduction in the proviral DNA (the 'reservoir'), in this 'proof-of-concept' study, in those randomised to the vaccine-HDACi intervention compared to those receiving antiretroviral therapy alone.

ELIGIBILITY:
Inclusion criteria

1. Aged ≥18 to ≤60 years old
2. Able to give informed written consent including consent to long-term follow-up
3. Should be enrolled within a maximum of 4 weeks of a diagnosis of primary HIV-1 infection confirmed by one of the following criteria:

   1. Positive HIV-1 serology within a maximum of 12 weeks of a documented negative HIV-1 serology test result (can include point of care test (POCT) using blood for both tests)
   2. A positive p24 antigen result and a negative HIV antibody test
   3. Negative antibody test with either detectable HIV RNA or proviral DNA
   4. PHE RITA test algorithm (a) reported as "Incident" confirming the HIV-1 antibody avidity is consistent with recent infection (within the preceding 16 weeks).
   5. Weakly reactive or equivocal 4th generation HIV antibody antigen test
   6. Equivocal or reactive antibody test with <4 bands on western blot
4. Adequate haemoglobin (Hb≥12g/dL for males, ≥11g/dL for females)
5. Weight ≥50kg
6. Willing to be treated with cART (preferably including raltegravir) and be randomised to continue cART alone or cART plus intervention (HIV vaccines plus HDACi)
7. Willing and able to comply with visit schedule and provide blood sampling

Exclusion criteria

1. Women of child bearing potential (WCBP) (b)
2. In women with intact ovaries and no uterus, any planned egg donation anytime in the future to a surrogate
3. Intention to donate sperm or father a child within 6 months of the intervention
4. Co-infection with hepatitis B (surface antigen positive or detectable HBV DNA levels in blood) or hepatitis C (HCV RNA positive or HVC antigen positive)
5. Any current or past history of malignancy
6. Concurrent opportunistic infection or other comorbidity or comorbidity likely to occur during the trial e.g.past history of ischaemic or other significant heart disease, malabsorption syndromes, autoimmune disease
7. Any contraindication to receipt of BHIVA recommended combination antiretrovirals
8. HIV-2 infection
9. Known HTLV-1 co-infection
10. Prior immunisation with any experimental HIV Immunogens (including any component of the vaccines used in the RIVER protocol; simian or human adenoviral vaccine; other experimental HIV vaccines)
11. Current or planned systemic immunosuppressive therapy (inhaled corticosteroids are allowed)
12. Any history of proven thromboembolism (pulmonary embolism or deep vein thrombosis)
13. Any inherited or acquired bleeding diathesis including gastric or duodenal ulcers, varices
14. Concurrent or planned use of any drugs contraindicated with vorinostat i.e. antiarrhythmics; any other drugs that prolong QTc; warfarin, aspirin, sodium valproate
15. Prior intolerance of any of either the components of the vaccine or HDACi,
16. Uncontrolled diabetes mellitus defined as an HBA1C>7%
17. Any congenital or acquired prolongation of the QTc interval, with normal defined as ≤0.44s (≤440ms)
18. Participation in any other clinical trial of an experimental agent or any non-interventional study where additional blood draws are required; participation in an observational study is permitted
19. Allergy to egg
20. History of anaphylaxis or severe adverse reaction to vaccines
21. Planned receipt of vaccines within 2 weeks of the first trial vaccination administered at PR week 00 (including vaccines such as yellow fever; hepatitis B, influenza)
22. Abnormal blood test results at screening including:

    1. Moderate to severe hepatic impairment as defined by Child-Pugh classification
    2. ALT >5xULN
    3. Platelets <150x109/L
    4. eGFR <60 (c)
    5. uPCR >30 mg/mmol
23. Physical and laboratory test findings: Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination and/or vital signs that the investigator believes is a preclusion from enrolment into the study
24. Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate adherence with study requirements
25. Insufficient venous access that will allow scheduled blood draws as per protocol

    1. using current cut-offs for optical density as defined by PHE
    2. females aged <20 years of age, and weighing <65kg and <168cm in height will need to have an estimation of blood volume (EBV) prior to enrolment, >3500mL before to participate. This circumstance is unlikely to arise as most women between the ages of 18 to 20 years would be of child-bearing potential (CBP) and excluded on that basis.
    3. eGFR is calculated by the local labs using CKD-EPI. Units ml/min/1.73m2.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fidler, MD, Principal Investigator — Imperial College London
Locations (6):
- United Kingdom (6):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Central and North West London NHS Foundation Trust, London
  - Chelsea and Westminster NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Royal Free Hospital NHS Foundation Trust, London

REFERENCES:
- [Background] International AIDS Society Scientific Working Group on HIV Cure; Deeks SG, Autran B, Berkhout B, Benkirane M, Cairns S, Chomont N, Chun TW, Churchill M, Di Mascio M, Katlama C, Lafeuillade A, Landay A, Lederman M, Lewin SR, Maldarelli F, Margolis D, Markowitz M, Martinez-Picado J, Mullins JI, Mellors J, Moreno S, O'Doherty U, Palmer S, Penicaud MC, Peterlin M, Poli G, Routy JP, Rouzioux C, Silvestri G, Stevenson M, Telenti A, Van Lint C, Verdin E, Woolfrey A, Zaia J, Barre-Sinoussi F. Towards an HIV cure: a global scientific strategy. Nat Rev Immunol. 2012 Jul 20;12(8):607-14. doi: 10.1038/nri3262. PMID 22814509
- [Background] Rasmussen TA, Schmeltz Sogaard O, Brinkmann C, Wightman F, Lewin SR, Melchjorsen J, Dinarello C, Ostergaard L, Tolstrup M. Comparison of HDAC inhibitors in clinical development: effect on HIV production in latently infected cells and T-cell activation. Hum Vaccin Immunother. 2013 May;9(5):993-1001. doi: 10.4161/hv.23800. Epub 2013 Jan 31. PMID 23370291
- [Background] Richman DD. Introduction: challenges to finding a cure for HIV infection. Curr Opin HIV AIDS. 2011 Jan;6(1):1-3. doi: 10.1097/COH.0b013e328340ffa6. PMID 21242886
- [Background] Bolden JE, Peart MJ, Johnstone RW. Anticancer activities of histone deacetylase inhibitors. Nat Rev Drug Discov. 2006 Sep;5(9):769-84. doi: 10.1038/nrd2133. PMID 16955068
- [Background] Archin NM, Cheema M, Parker D, Wiegand A, Bosch RJ, Coffin JM, Eron J, Cohen M, Margolis DM. Antiretroviral intensification and valproic acid lack sustained effect on residual HIV-1 viremia or resting CD4+ cell infection. PLoS One. 2010 Feb 23;5(2):e9390. doi: 10.1371/journal.pone.0009390. PMID 20186346
- [Background] Contreras X, Schweneker M, Chen CS, McCune JM, Deeks SG, Martin J, Peterlin BM. Suberoylanilide hydroxamic acid reactivates HIV from latently infected cells. J Biol Chem. 2009 Mar 13;284(11):6782-9. doi: 10.1074/jbc.M807898200. Epub 2009 Jan 9. PMID 19136668
- [Background] Archin NM, Espeseth A, Parker D, Cheema M, Hazuda D, Margolis DM. Expression of latent HIV induced by the potent HDAC inhibitor suberoylanilide hydroxamic acid. AIDS Res Hum Retroviruses. 2009 Feb;25(2):207-12. doi: 10.1089/aid.2008.0191. PMID 19239360
- [Background] Archin NM, Vaidya NK, Kuruc JD, Liberty AL, Wiegand A, Kearney MF, Cohen MS, Coffin JM, Bosch RJ, Gay CL, Eron JJ, Margolis DM, Perelson AS. Immediate antiviral therapy appears to restrict resting CD4+ cell HIV-1 infection without accelerating the decay of latent infection. Proc Natl Acad Sci U S A. 2012 Jun 12;109(24):9523-8. doi: 10.1073/pnas.1120248109. Epub 2012 May 29. PMID 22645358
- [Background] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Background] Shan L, Deng K, Shroff NS, Durand CM, Rabi SA, Yang HC, Zhang H, Margolick JB, Blankson JN, Siliciano RF. Stimulation of HIV-1-specific cytolytic T lymphocytes facilitates elimination of latent viral reservoir after virus reactivation. Immunity. 2012 Mar 23;36(3):491-501. doi: 10.1016/j.immuni.2012.01.014. Epub 2012 Mar 8. PMID 22406268
- [Background] Letourneau S, Im EJ, Mashishi T, Brereton C, Bridgeman A, Yang H, Dorrell L, Dong T, Korber B, McMichael AJ, Hanke T. Design and pre-clinical evaluation of a universal HIV-1 vaccine. PLoS One. 2007 Oct 3;2(10):e984. doi: 10.1371/journal.pone.0000984. PMID 17912361
- [Background] Rollier CS, Reyes-Sandoval A, Cottingham MG, Ewer K, Hill AV. Viral vectors as vaccine platforms: deployment in sight. Curr Opin Immunol. 2011 Jun;23(3):377-82. doi: 10.1016/j.coi.2011.03.006. Epub 2011 Apr 20. PMID 21514130
- [Background] Kostense S, Koudstaal W, Sprangers M, Weverling GJ, Penders G, Helmus N, Vogels R, Bakker M, Berkhout B, Havenga M, Goudsmit J. Adenovirus types 5 and 35 seroprevalence in AIDS risk groups supports type 35 as a vaccine vector. AIDS. 2004 May 21;18(8):1213-6. doi: 10.1097/00002030-200405210-00019. PMID 15166541
- [Background] Tatsis N, Blejer A, Lasaro MO, Hensley SE, Cun A, Tesema L, Li Y, Gao GP, Xiang ZQ, Zhou D, Wilson JM, Ertl HC. A CD46-binding chimpanzee adenovirus vector as a vaccine carrier. Mol Ther. 2007 Mar;15(3):608-17. doi: 10.1038/sj.mt.6300078. Epub 2007 Jan 16. PMID 17228314
- [Background] Colloca S, Barnes E, Folgori A, Ammendola V, Capone S, Cirillo A, Siani L, Naddeo M, Grazioli F, Esposito ML, Ambrosio M, Sparacino A, Bartiromo M, Meola A, Smith K, Kurioka A, O'Hara GA, Ewer KJ, Anagnostou N, Bliss C, Hill AV, Traboni C, Klenerman P, Cortese R, Nicosia A. Vaccine vectors derived from a large collection of simian adenoviruses induce potent cellular immunity across multiple species. Sci Transl Med. 2012 Jan 4;4(115):115ra2. doi: 10.1126/scitranslmed.3002925. PMID 22218691
- [Background] Barnes E, Folgori A, Capone S, Swadling L, Aston S, Kurioka A, Meyer J, Huddart R, Smith K, Townsend R, Brown A, Antrobus R, Ammendola V, Naddeo M, O'Hara G, Willberg C, Harrison A, Grazioli F, Esposito ML, Siani L, Traboni C, Oo Y, Adams D, Hill A, Colloca S, Nicosia A, Cortese R, Klenerman P. Novel adenovirus-based vaccines induce broad and sustained T cell responses to HCV in man. Sci Transl Med. 2012 Jan 4;4(115):115ra1. doi: 10.1126/scitranslmed.3003155. PMID 22218690
- [Background] Sheehy SH, Duncan CJ, Elias SC, Collins KA, Ewer KJ, Spencer AJ, Williams AR, Halstead FD, Moretz SE, Miura K, Epp C, Dicks MD, Poulton ID, Lawrie AM, Berrie E, Moyle S, Long CA, Colloca S, Cortese R, Gilbert SC, Nicosia A, Hill AV, Draper SJ. Phase Ia clinical evaluation of the Plasmodium falciparum blood-stage antigen MSP1 in ChAd63 and MVA vaccine vectors. Mol Ther. 2011 Dec;19(12):2269-76. doi: 10.1038/mt.2011.176. Epub 2011 Aug 23. PMID 21862998
- [Background] Mayr A, Stickl H, Muller HK, Danner K, Singer H. [The smallpox vaccination strain MVA: marker, genetic structure, experience gained with the parenteral vaccination and behavior in organisms with a debilitated defence mechanism (author's transl)]. Zentralbl Bakteriol B. 1978 Dec;167(5-6):375-90. German. PMID 219640
- [Background] Drexler I, Heller K, Wahren B, Erfle V, Sutter G. Highly attenuated modified vaccinia virus Ankara replicates in baby hamster kidney cells, a potential host for virus propagation, but not in various human transformed and primary cells. J Gen Virol. 1998 Feb;79 ( Pt 2):347-52. doi: 10.1099/0022-1317-79-2-347. PMID 9472619
- [Background] Sutter G, Moss B. Nonreplicating vaccinia vector efficiently expresses recombinant genes. Proc Natl Acad Sci U S A. 1992 Nov 15;89(22):10847-51. doi: 10.1073/pnas.89.22.10847. PMID 1438287
- [Background] Hanke T, Samuel RV, Blanchard TJ, Neumann VC, Allen TM, Boyson JE, Sharpe SA, Cook N, Smith GL, Watkins DI, Cranage MP, McMichael AJ. Effective induction of simian immunodeficiency virus-specific cytotoxic T lymphocytes in macaques by using a multiepitope gene and DNA prime-modified vaccinia virus Ankara boost vaccination regimen. J Virol. 1999 Sep;73(9):7524-32. doi: 10.1128/JVI.73.9.7524-7532.1999. PMID 10438842
- [Background] Schmitz JE, Kuroda MJ, Santra S, Sasseville VG, Simon MA, Lifton MA, Racz P, Tenner-Racz K, Dalesandro M, Scallon BJ, Ghrayeb J, Forman MA, Montefiori DC, Rieber EP, Letvin NL, Reimann KA. Control of viremia in simian immunodeficiency virus infection by CD8+ lymphocytes. Science. 1999 Feb 5;283(5403):857-60. doi: 10.1126/science.283.5403.857. PMID 9933172
- [Background] Barouch DH, Santra S, Kuroda MJ, Schmitz JE, Plishka R, Buckler-White A, Gaitan AE, Zin R, Nam JH, Wyatt LS, Lifton MA, Nickerson CE, Moss B, Montefiori DC, Hirsch VM, Letvin NL. Reduction of simian-human immunodeficiency virus 89.6P viremia in rhesus monkeys by recombinant modified vaccinia virus Ankara vaccination. J Virol. 2001 Jun;75(11):5151-8. doi: 10.1128/JVI.75.11.5151-5158.2001. PMID 11333896
- [Background] Hayton EJ, Rose A, Ibrahimsa U, Del Sorbo M, Capone S, Crook A, Black AP, Dorrell L, Hanke T. Safety and tolerability of conserved region vaccines vectored by plasmid DNA, simian adenovirus and modified vaccinia virus ankara administered to human immunodeficiency virus type 1-uninfected adults in a randomized, single-blind phase I trial. PLoS One. 2014 Jul 9;9(7):e101591. doi: 10.1371/journal.pone.0101591. eCollection 2014. PMID 25007091
- [Background] Kinloch-de Loes S, Hoen B, Smith DE, Autran B, Lampe FC, Phillips AN, Goh LE, Andersson J, Tsoukas C, Sonnerborg A, Tambussi G, Girard PM, Bloch M, Battegay M, Carter N, El Habib R, Theofan G, Cooper DA, Perrin L; QUEST Study Group. Impact of therapeutic immunization on HIV-1 viremia after discontinuation of antiretroviral therapy initiated during acute infection. J Infect Dis. 2005 Aug 15;192(4):607-17. doi: 10.1086/432002. Epub 2005 Jul 15. PMID 16028129
- [Background] Vanham G, Van Gulck E. Can immunotherapy be useful as a "functional cure" for infection with Human Immunodeficiency Virus-1? Retrovirology. 2012 Sep 7;9:72. doi: 10.1186/1742-4690-9-72. PMID 22958464
- [Background] Dorrell L, Yang H, Ondondo B, Dong T, di Gleria K, Suttill A, Conlon C, Brown D, Williams P, Bowness P, Goonetilleke N, Rostron T, Rowland-Jones S, Hanke T, McMichael A. Expansion and diversification of virus-specific T cells following immunization of human immunodeficiency virus type 1 (HIV-1)-infected individuals with a recombinant modified vaccinia virus Ankara/HIV-1 Gag vaccine. J Virol. 2006 May;80(10):4705-16. doi: 10.1128/JVI.80.10.4705-4716.2006. PMID 16641264
- [Background] Hicks CB, Gay C, Ferrari G. Acute HIV infection: the impact of anti-retroviral treatment on cellular immune responses. Clin Exp Immunol. 2007 Aug;149(2):211-6. doi: 10.1111/j.1365-2249.2007.03437.x. Epub 2007 Jun 21. PMID 17590167
- [Background] Evering TH, Mehandru S, Racz P, Tenner-Racz K, Poles MA, Figueroa A, Mohri H, Markowitz M. Absence of HIV-1 evolution in the gut-associated lymphoid tissue from patients on combination antiviral therapy initiated during primary infection. PLoS Pathog. 2012 Feb;8(2):e1002506. doi: 10.1371/journal.ppat.1002506. Epub 2012 Feb 2. PMID 22319447
- [Background] Goujard C, Girault I, Rouzioux C, Lecuroux C, Deveau C, Chaix ML, Jacomet C, Talamali A, Delfraissy JF, Venet A, Meyer L, Sinet M; ANRS CO6 PRIMO Study Group. HIV-1 control after transient antiretroviral treatment initiated in primary infection: role of patient characteristics and effect of therapy. Antivir Ther. 2012;17(6):1001-9. doi: 10.3851/IMP2273. Epub 2012 Aug 6. PMID 22865544
- [Background] SPARTAC Trial Investigators; Fidler S, Porter K, Ewings F, Frater J, Ramjee G, Cooper D, Rees H, Fisher M, Schechter M, Kaleebu P, Tambussi G, Kinloch S, Miro JM, Kelleher A, McClure M, Kaye S, Gabriel M, Phillips R, Weber J, Babiker A. Short-course antiretroviral therapy in primary HIV infection. N Engl J Med. 2013 Jan 17;368(3):207-17. doi: 10.1056/NEJMoa1110039. PMID 23323897
- [Background] Ngo-Giang-Huong N, Deveau C, Da Silva I, Pellegrin I, Venet A, Harzic M, Sinet M, Delfraissy JF, Meyer L, Goujard C, Rouzioux C; Frnech PRIMO Cohort Study Group. Proviral HIV-1 DNA in subjects followed since primary HIV-1 infection who suppress plasma viral load after one year of highly active antiretroviral therapy. AIDS. 2001 Apr 13;15(6):665-73. doi: 10.1097/00002030-200104130-00001. PMID 11371680
- [Background] Koelsch KK, Boesecke C, McBride K, Gelgor L, Fahey P, Natarajan V, Baker D, Bloch M, Murray JM, Zaunders J, Emery S, Cooper DA, Kelleher AD; PINT study team. Impact of treatment with raltegravir during primary or chronic HIV infection on RNA decay characteristics and the HIV viral reservoir. AIDS. 2011 Nov 13;25(17):2069-78. doi: 10.1097/QAD.0b013e32834b9658. PMID 21860347
- [Result] Hamlyn E, Ewings FM, Porter K, Cooper DA, Tambussi G, Schechter M, Pedersen C, Okulicz JF, McClure M, Babiker A, Weber J, Fidler S; INSIGHT SMART and SPARTAC Investigators. Plasma HIV viral rebound following protocol-indicated cessation of ART commenced in primary and chronic HIV infection. PLoS One. 2012;7(8):e43754. doi: 10.1371/journal.pone.0043754. Epub 2012 Aug 31. PMID 22952756
- [Result] Eisele E, Siliciano RF. Redefining the viral reservoirs that prevent HIV-1 eradication. Immunity. 2012 Sep 21;37(3):377-88. doi: 10.1016/j.immuni.2012.08.010. PMID 22999944
- [Result] Coiras M, Lopez-Huertas MR, Perez-Olmeda M, Alcami J. Understanding HIV-1 latency provides clues for the eradication of long-term reservoirs. Nat Rev Microbiol. 2009 Nov;7(11):798-812. doi: 10.1038/nrmicro2223. PMID 19834480
- [Result] Chun TW, Fauci AS. HIV reservoirs: pathogenesis and obstacles to viral eradication and cure. AIDS. 2012 Jun 19;26(10):1261-8. doi: 10.1097/QAD.0b013e328353f3f1. PMID 22472858
- [Result] Archin NM, Keedy KS, Espeseth A, Dang H, Hazuda DJ, Margolis DM. Expression of latent human immunodeficiency type 1 is induced by novel and selective histone deacetylase inhibitors. AIDS. 2009 Sep 10;23(14):1799-806. doi: 10.1097/QAD.0b013e32832ec1dc. PMID 19590405
- [Result] Hutter G, Nowak D, Mossner M, Ganepola S, Mussig A, Allers K, Schneider T, Hofmann J, Kucherer C, Blau O, Blau IW, Hofmann WK, Thiel E. Long-term control of HIV by CCR5 Delta32/Delta32 stem-cell transplantation. N Engl J Med. 2009 Feb 12;360(7):692-8. doi: 10.1056/NEJMoa0802905. PMID 19213682
- [Result] Saez-Cirion A, Bacchus C, Hocqueloux L, Avettand-Fenoel V, Girault I, Lecuroux C, Potard V, Versmisse P, Melard A, Prazuck T, Descours B, Guergnon J, Viard JP, Boufassa F, Lambotte O, Goujard C, Meyer L, Costagliola D, Venet A, Pancino G, Autran B, Rouzioux C; ANRS VISCONTI Study Group. Post-treatment HIV-1 controllers with a long-term virological remission after the interruption of early initiated antiretroviral therapy ANRS VISCONTI Study. PLoS Pathog. 2013 Mar;9(3):e1003211. doi: 10.1371/journal.ppat.1003211. Epub 2013 Mar 14. PMID 23516360
- [Result] Deeks SG. HIV: Shock and kill. Nature. 2012 Jul 25;487(7408):439-40. doi: 10.1038/487439a. No abstract available. PMID 22836995
- [Result] Fidler S, Stohr W, Pace M, Dorrell L, Lever A, Pett S, Kinloch-de Loes S, Fox J, Clarke A, Nelson M, Thornhill J, Khan M, Fun A, Bandara M, Kelly D, Kopycinski J, Hanke T, Yang H, Bennett R, Johnson M, Howell B, Barnard R, Wu G, Kaye S, Wills M, Babiker A, Frater J; RIVER trial study group. Antiretroviral therapy alone versus antiretroviral therapy with a kick and kill approach, on measures of the HIV reservoir in participants with recent HIV infection (the RIVER trial): a phase 2, randomised trial. Lancet. 2020 Mar 14;395(10227):888-898. doi: 10.1016/S0140-6736(19)32990-3. Epub 2020 Feb 19. PMID 32085823
- See also: CHERUB (Collaborative HIV Eradication of viral Reservoirs: UK BRC) website — http://www.cherub.uk.net/
- See also: Medical Research Council Clinical Trials Unit — http://www.ctu.mrc.ac.uk/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 UK clinical sites. The recruitment period was from November 2015 until July 2017. Last patient last visit was completed in November 2017.
Pre-assignment Details: Participants were recruited from two Strata:
  1. Recently diagnosed with primary HIV-1 infection - Eligible participants were enrolled at week 0 when combination ART (cART) began. Randomisation occurred at week 22
  2. Previously diagnosed with primary HIV-1 infection - Randomisation occurred within 2 weeks of screening.
Groups:
- Control: Participants received combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed for the duration of the study
- Intervention: Participants received combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed for the duration of the study Plus ChAdV63.HIVconsv prime (post-randomisation week 00) and MVA.HIVconsv boost (post randomisation week 08 day 1) vaccines; followed by a 28-day course of vorinostat (10 doses in total).
Period: Overall Study
Arm/Group | Control | Intervention
Started | 30 | 30
Completed | 30 | 28
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control (Arm A - ART Only): Combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed at week 0 for the duration of the study up to post-randomisation week 18 (42 weeks in total)
- Intervention (Arm B - ART + Vaccines + Vorinostat): Combination Antiretroviral Therapy (cART) preferably including raltegravir prescribed at week 0 for the duration of the study up to post-randomisation week 18 (42 weeks in total) Plus ChAdV63.HIVconsv prime (post-randomisation week 00) and MVA.HIVconsv boost (post randomisation week 08 day 1) vaccines; followed by a 28-day course of vorinostat (10 doses in total).
- Total: Total of all reporting groups
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [30 to 38] | 35 [28 to 44] | 32 [29 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 26 | 42
  South Asian | 0 | 1 | 1
  South East Asian | 1 | 0 | 1
  Hispanic/Latino | 3 | 2 | 5
  Black Caribbean/American | 2 | 0 | 2
  Black African | 2 | 0 | 2
  Mixed ethnic group | 5 | 1 | 6
  Other | 1 | 0 | 1
Mode of HIV Infection [Count of Participants; unit: Participants] — MSM = men who have sex with men MSW = men who have sex with women IDU = Injection Drug Use
  Participants
    MSM | 26 | 29 | 55
    MSW | 1 | 1 | 2
    MSM + IDU | 2 | 0 | 2
    Unknown | 1 | 0 | 1
CD4 at randomisation [Median (Inter-Quartile Range); unit: cells/mm3] | 694 [561 to 844] | 710 [579 to 759] | 708 [568 to 788]
HIV RNA at randomisation (copies/ml) [Count of Participants; unit: Participants]
  <50 | 29 | 30 | 59
  50 - <200 | 1 | 0 | 1
Weeks since PHI diagnosis [Count of Participants; unit: Participants] — PHI = Primary HIV Infection
  Participants
    <= 1 week | 1 | 0 | 1
    >1 - 2 weeks | 3 | 3 | 6
    >2 - 3 weeks | 7 | 7 | 14
    >3 - 4 weeks | 15 | 16 | 31
    > 4 weeks | 4 | 4 | 8
Weeks since PHI diagnosis (at randomisation) [Median (Inter-Quartile Range); unit: weeks] | 28 [27 to 41] | 28 [27 to 34] | 28 [27 to 36]

OUTCOME MEASURES:

1. Primary Outcome: Total HIV DNA From CD4 T-cells
Description: The average of two measures taken at post-randomisation week 16 and 18
Time Frame: Averaged across post-randomisation week 16 and 18
Measure: Mean (Standard Deviation); unit: HIV-DNA copies/mill CD4+ T cells (log10)
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 30 | 30
HIV-DNA copies/mill CD4+ T cells (log10) | 2.95 (0.50) | 3.06 (0.49)
Statistical Analysis 1: Comparison: Control (Arm A - ART Only) vs Intervention (Arm B - ART + Vaccines + Vorinostat); Test type: Superiority; p = 0.26, Regression, Linear — Treatment arms were compared in terms of absolute total HIV DNA levels (on a log10-scale) at post-randomization weeks 16 and 18 adjusted for the baseline (i.e. randomization) level and by stratum

2. Secondary Outcome: Clinical Adverse Events
Description: Clinical adverse events of any grade post-randomization.
Time Frame: From randomization to the final visit at week 18.
Population: All participants randomized
Measure: Count of Participants; unit: Participants
Groups:
- Control (Arm A - ART Only): Combination Antiretroviral Therapy (cART): Likely consisting of an Nucleoside reverse-transcriptase inhibitor (NRTI) backbone i.e. Truvada plus a ritonavir-boosted protease inhibitor (PI) e.g. Darunavir + ritonavir. Prescribed at week 0 for the duration of the study.
  Raltegravir: All participants will be dispensed sufficient supplies of Raltegravir to ensure they have sufficient medication to last to the next study visit. Raltegravir is supplied in marketed pack with 30 tablets per bottle.
- Intervention (Arm B - ART + Vaccines + Vorinostat): ART plus vaccines plus vorinostat
  Combination Antiretroviral Therapy (cART): Likely consisting of an Nucleoside reverse-transcriptase inhibitor (NRTI) backbone i.e. Truvada plus a ritonavir-boosted protease inhibitor (PI) e.g. Darunavir + ritonavir. Prescribed at week 0 for the duration of the study.
  Raltegravir: All participants will be dispensed sufficient supplies of Raltegravir to ensure they have sufficient medication to last to the next study visit. Raltegravir is supplied in marketed pack with 30 tablets per bottle.
  Vorinostat: Vorinostat (suberoylanilide hydroxamic acid abbreviated to SAHA) inhibits the histone deacetylases HDAC1, HDAC2, HDA
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 30 | 30
Participants
  Not had any event | 8 | 1
  Did have any event | 22 | 29

3. Secondary Outcome: Quantitative Viral Outgrowth
Description: Number of Participants with undetectable quantitative viral outgrowth
Time Frame: At week 16
Population: All participants randomized with valid assay results at week 16.
Measure: Number; unit: Participants with undetectable outgrowth
Groups:
- Control (Arm A - ART Only): ART only
  Combination Antiretroviral Therapy (cART): Likely consisting of an Nucleoside reverse-transcriptase inhibitor (NRTI) backbone i.e. Truvada plus a ritonavir-boosted protease inhibitor (PI) e.g. Darunavir + ritonavir. Prescribed at week 0 for the duration of the study.
  Raltegravir: All participants will be dispensed sufficient supplies of Raltegravir to ensure they have sufficient medication to last to the next study visit. Raltegravir is supplied in marketed pack with 30 tablets per bottle.
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 29 | 27
Participants with undetectable outgrowth | 12 | 6
Statistical Analysis 1: Comparison: Control (Arm A - ART Only) vs Intervention (Arm B - ART + Vaccines + Vorinostat); Comparison of the proportion of patients with undetectable viral outgrowth using logistic regression. The analysis was adjusted for stratum and baseline viral outgrowth. Missing baseline values were imputed; Test type: Superiority; p = 0.145, Regression, Logistic; Odds Ratio (OR) = 0.41

4. Secondary Outcome: Percentage of CD4+ CD154+ IFNγ+ T Cells
Description: Percentage of CD4+ CD154+ IFNγ+ T cells , assessed using an optimized and qualified flow cytometry panel.
Time Frame: 12 weeks
Population: All participants randomized with valid assay results
Measure: Median (Inter-Quartile Range); unit: % cells CD4+ CD154+ IFNγ+
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 27 | 30
% cells CD4+ CD154+ IFNγ+
  Post randomisation week 9 | 0.006 [0.000 to 0.015] | 0.097 [0.043 to 0.161]
  Post randomisation week 12 | 0.006 [0.000 to 0.015] | 0.109 [0.050 to 0.214]

5. Secondary Outcome: CD8+ T-cell Responses
Description: Percentage of CD8+ CD107a+ IFNγ+ T cells , assessed using an optimized and qualified flow cytometry panel.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: % cells CD8+ CD107a+ IFNγ+
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 27 | 30
% cells CD8+ CD107a+ IFNγ+
  Post randomisation week 9 | 0.052 [0.014 to 0.142] | 0.194 [0.142 to 0.722]
  Post randomisation week 12 | 0.062 [0.008 to 0.106] | 0.263 [0.105 to 0.620]

6. Secondary Outcome: Viral Inhibition
Description: CD8+ T cell antiviral suppressive activity was expressed as percentage elimination and determined as follows: [(fraction of p24+ cells in CD4+ T cells cultured alone) - (fraction of p24 + in CD4+ T cells cultured with CD8+ cells)]/(fraction of p24+ cells in CD4+ T cells cultured alone) × 100.
  Viral inhibition Assay
Time Frame: 12 weeks
Population: All participants randomized with valid assay results
Measure: Mean (95% Confidence Interval); unit: Percentage elimination
Groups:
- Control (Arm A - ART Only): ART only
  Raltegravir: All participants will be dispensed sufficient supplies of Raltegravir to ensure they have sufficient medication to last to the next study visit. Raltegravir is supplied in marketed pack with 30 tablets per bottle.
Arm/Group | Control (Arm A - ART Only) | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 27 | 30
Percentage elimination | -18.25 [-29.65 to -6.85] | 1.50 [-11.28 to 14.27]

7. Post Hoc Outcome: Histone H4 Acetylation
Description: Histone H4 acetylation using a H4K5/8/12/16 immunoassay with thawed PBMC derived cell lysates added to an ELISA using anti-H4 monoclonal antibody
Time Frame: 12 weeks
Population: Intervention arm only - histone H4 acetylation was only measured in participants in the intervention arm with the aim to compare values approximately 2 hours post vorinostat intake with values pre vorinostat intake. No data were collected from participants in the control arm.
Measure: Mean (95% Confidence Interval); unit: Fold increase pre to post vorinostat
Arm/Group | Intervention (Arm B - ART + Vaccines + Vorinostat)
Number analyzed (Participants) | 22
Fold increase pre to post vorinostat | 3.19 [2.42 to 4.22]

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- Control: ART only
  Combination ART (cART) preferably including raltegravir (control)
- Intervention: ART plus vaccines plus vorinostat
  Combination ART (cART) preferably including raltegravir* plus ChAdV63.HIVconsv (ChAd) prime and MVA.HIVconsv (MVA) boost vaccines; followed by a 28-day course of vorinostat (10 doses in total).
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/30
Other Adverse Events (participants affected / at risk) | 6/30 | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=30) | Intervention (N=30)
Vasovagal syncope (Vascular disorders) | 0 (0) | 1 (1) — Vasovagal syncope likely secondary to venesection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=30) | Intervention (N=30)
Acute hepatitis A (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3 hepatitis
Influenza (Infections and infestations) | 1 (1) | 0 (0) — Grade 3 influenza
Proctitis herpes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 3 proctitis herpes
Shingles (Infections and infestations) | 1 (1) | 0 (0) — Grade 3 shingles
Wrist injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 3 wrist injury
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) — Grade 3 back pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The NHS Organisations shall not publish or otherwise disseminate conclusions of the Study, including all or any part of the Results of the Study without prior written consent of the Sponsor, such consent not to be unreasonably withheld or delayed.

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT02336074/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT02336074/SAP_001.pdf